CLINICAL TRIAL: NCT05350189
Title: GUS: Gadavist Drug Utilization Study
Brief Title: A Study Called GUS to Understand How Much of the Contrast Agent Gadavist is Used and How Much is Wasted in Two Different Containers (Single-dose Vials and Imaging Bulk Packages ) in a Real-world Setting
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22072
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Contrast Enhancement in Magnetic Resonance Imaging
MeSH Terms: interventions — gadobutrol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Gadavist Single-dose vial: Data will be collected from contrast-enhanced Magnetic Resonance Imaging (MRI) using Gadavist from a single-dose vial of 7.5 or 10 or 15 milliliters (mL).
  Interventions: Drug: Gadobutrol (Gadavist/Gadovist, BAY86-4875)
- Gadavist IBP: Data will be collected from contrast-enhanced MRI using Gadavist from an IBP of either 30 or 65 milliliters (mL), and from Gadavist via a single-dose vial due to insufficient product remaining in an IBP during the IBP cohort.
  Interventions: Drug: Gadobutrol (Gadavist/Gadovist, BAY86-4875)

INTERVENTIONS:
Drug: Gadobutrol (Gadavist/Gadovist, BAY86-4875) — At discretion of attending physician

SUMMARY:
This is an observational study, in which data associated with the wastage with the use of Gadavist single-dose vials, as compared to the wastage associated with the use of the Gadavist imaging bulk packages (IBP) used for contrast-enhanced magnetic resonance imaging (MRI) using Gadavist will be compared.

MRI is a medical technique, which creates detailed images of the organs, soft tissues and structures inside the body. Combination of MRI with a "dye" that is injected into the vein (called contrast media, like Gadavist) creates what is called a contrast-enhanced MRI that enables clearer pictures of the body and helps doctors to see problems better than an MRI without contrast media.

The drug Gadavist (also called gadobutrol) is a gadolinium-based contrast media for diagnostic use in MRI, which is given as an injection into the vein to improve the quality of the MRI pictures. Gadavist is already approved for several indications including imaging of brain and spinal cord, breast imaging, imaging of blood vessels, and diagnoses of heart disease. It helps doctors for example to detect:

* areas with disrupted blood brain barrier (BBB), which is crucial to protect the brain from toxic components and pathogens (germs, viruses, disease-causing agents)
* abnormal blood vessels in certain blood vessels
* presence and size of breast cancer
* heart disease The dosing of Gadavist is weight-based and currently available in single-use vials, which are associated with wastage. To reduce wastage and wastage associated costs, multi-dose vials, also called imaging bulk packages (IBP) were developed, which are already approved in the USA since January 2021.

The aim of this study is to understand how much of the contrast agent Gadavist is used and how much is wasted in two different containers (single-dose vials and Imaging Bulk Packages (IBP)) in a real-world setting. To do this, researchers will review information collected regarding the amount of Gadavist used for patients undergoing contrast-enhanced MRI for any indication regarding:

* vial type (single-dose or IBP)
* size of single-dose or IBP
* volume of administered dose (mL)
* date of administration
* time of administration
* injection modality (manual vs power)
* type of power injector, if applicable

There will be no study-mandated visits or treatments. The decision to undergo a contrast-enhanced MRI with Gadavist will be made by the study participants with their doctors before data collection, and independently of this study. Data will be collected over a period of approximately 6-weeks, until the data collection of 1200 participants for each comparison group (vial type) is completed. No patient information beyond Gadavist dose will be collected in this study.

ELIGIBILITY:
Inclusion Criteria:

* A contrast-enhanced MRI using Gadavist for any indication at the study site during the study period
* Scheduled MRI to be performed in a study-designated room

Exclusion Criteria:

* Administration of Gadavist from a single-dose prefilled syringe
* MRIs performed in the emergency setting

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes all contrast-enhanced non-emergency Magnetic Resonance Imaging (MRI) using Gadavist for any indication at the participating site during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 1602 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Overall total wastage in milliliter (mL) for single-dose vials consumed in the single-dose vial cohort | Up to 12 weeks
  Wastage will be defined as:
  For single-dose vials, any unused product that remains immediately following the administration of Gadavist to a single patient.
Overall total wastage in mL for IBPs and single-dose vials consumed in the IBP cohort | Up to 12 weeks
  Wastage will be defined as:
  For IBPs, any unused product that remains after the administration of Gadavist to some number of patients and where the allowable 24-hour window has expired, or in the event of office closure, would expire before the next scheduled Gadavist-enhanced MRI. Should a patient receive Gadavist via a single-dose vial due to insufficient product remaining in an IBP during the IBP cohort, the wastage from this single-dose vial will contribute to the overall wastage of that IBP.

SECONDARY OUTCOMES:
The cost associated with discarded Gadavist using the total volume of wastage for single-dose vials and IBPs cohort | Up to 12 weeks
The accuracy of the Bayer Radiology IBP cost calculator by comparing the estimated cost associated with discarded Gadavist as generated from the study analysis with the cost generated by the cost calculator | Up to 12 weeks
The average number of Gadavist administrations from each of the IBP volumes as assessed by administration counts recorded for each IBP vial sizes | Up to 12 weeks
The average dose of Gadavist administered from each of the IBP vial sizes as assessed by doses recorded for each IBP vial sizes | Up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.